

## **Non-Interventional Study Protocol**

| BI Study No.: | 1218.104 | | | |
|---|---|---|---|---|
| BI Investigational Product(s): | Linagliptin | | | |
| Title: | and effective | eness of Ti | nent non interventional study to monitor the safety<br>Trajenta ( <b>Lina</b> gliptin, 5 mg, q.d) in Korean<br>iabetes mellitus | у |
| | (SELINA s | tudy) | | |
| Clinical Phase: | IV | | | , |
| Trial Clinical<br>Monitor: | | | | |
| | Phone: | | Fax: | |
| Principal<br>Investigator: | Not Applica | able | | |
| Status: | Final protocol (Revised protocol) | | | |
| Version and Date: | Version: | 2.1 | <b>Date: 22 Feb 2017</b> | |
| Proprietary confidential information. | | | v4 | |

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

BI Trial No.: 1218.104

Doc. No.: UXX-XXX 

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## NON-INTERVENTIONAL STUDY PROTOCOL SYNOPSIS

| Name of company/Marketing Authorisation Holder: | | Tabulated<br>Study Protocol | |
|---|---|---|---|
| Boehringer Ingelheim Korea | | | |
| Name of finished produ | ict: | | |
| Trajenta | | | |
| Name of active ingredic | ent: | | |
| Linagliptin | | | |
| Protocol date: | Trial number: | | Revision date: |
| 1 December 2011 | 1218.104/UXX-<br>XXXX | | 22 Feb 2017 |
| Title of study: | | t non interventional study to monito<br>( <b>Lina</b> gliptin, 5 mg, q.d) in Korean<br>NA study) | |
| Principal<br>Investigator: | To be decided | | |
| Study site(s): | Multi-centre study | | |
| Clinical phase: | IV | | |
| | | ofile and effectiveness of linaglipting in a routine clinical practice setting | in Korean patients with |
| Methodology: Prospective, non-interven | | ntional, open-label, multi-centre nat | tional study |
| No. of patients: | | | |
| Total entered: | 3,000 approximately | | |
| each treatment: | Single arm (N=3,000 app | proximately) | |
| Diagnosis: | Patients diagnosed with | type 2 diabetes mellitus | |
| Main criteria for inclusion: | <ol> <li>No previous exposure to Trajenta</li> <li>Patients who have been started on Trajenta in accordance with the approved label in Korea</li> <li>No current participation in clinical trials</li> <li>Patients who have signed on the data release consent form</li> </ol> | | |
| Test product(s): | Linagliptin | | |
| dose: | 5 mg q.d | | |
| mode of admin. : | mode of admin.: Oral administration | | |
| Comparator product(s) | : Not applicable | | |
| dose: | | | |
| mode of admin. : | | | |

22 Feb 2017


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| Name of company/Marketing Authorisation Holder: | | Tabulated<br>Study Protocol | |
|---|---|---|---|
| Boehringer Ingelheim K | orea | | |
| Name of finished produ | ict: | | |
| Trajenta | | | |
| Name of active ingredie | ent: | | |
| Linagliptin | | | |
| Protocol date:<br>1 December 2011 | Trial number:<br>1218.104/UXX-<br>XXXX | | Revision date:<br>22 Feb 2017 |
| Duration of treatment: | 1) Treatment duration for short-term surveillance: 12±2 weeks, long-term surveillance: 24±2 weeks. 2) Study duration: 6 years. (KFDA set Trajenta re-examination period from 14 Sep 2011 to 13 Sep 2017. Interim report planned biannually for the initial two years | | |
| | and annually thereafter by Dec 2017.) | | |
| Criteria for effectiveness: | <ol> <li>Main endpoint</li> <li>Change from baseline in HbA1c after 24 weeks of treatment.</li> <li>Other endpoint</li> </ol> | | |
| | | to target effectiveness response, that after 24 weeks of treatment. | at is an HbA1c under |
| | 2) Occurrence of relative effectiveness response (HbA <sub>1c</sub> lowering by at least 0.5% after 24 weeks) | | |
| | 3) Change from baseline in fasting plasma glucose (FPG) after 24 weeks of treatment | | |
| Criteria for safety: | All reported adverse events including hypoglycemic events in patients who take at least one dose of Trajenta will be noted. | | |
| | Endpoints pertaining to safety will be presented as incidence rates of adverse events | | |
| Statistical methods: | s: Descriptive statistics | | |

**** 

Doc. No.: UXX-XXX Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## **FLOW CHART**

| Data points | Baseline | Follow-up 1 | Follow-up 2 |
|---|---|---|---|
| Visit Number | 1 | 2 | 3 |
| Week/s | 0 | 12±2 | 24±2 |
| Diagnosis | X | | |
| Inclusion / exclusion criteria | X | | |
| Demographics | X | | |
| Diabetes mellitus complications | X | | |
| Other medical history | X | | |
| Anti-hyperglycemic agents | X | X | X |
| Concomitant medications | X | X | X |
| Trajenta administration status | X | X | X |
| Renal function | X <sup>A</sup> | | |
| Effectiveness endpoints | X | X | X |
| Changes in lab tests | | X <sup>A</sup> | X <sup>A</sup> |
| Adverse events | | X | X |
| Study completion | | X | X |

A: If applicable.

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## **TABLE OF CONTENTS**

| TIT | LE 1 | PAGE | 오류! 책갈피가 정의되어 있지 않습! | 니다. |
|---|---|---|---|---|
| NO | N-IN | TERV | VENTIONAL STUDY PROTOCOL SYNOPSIS | 2 |
| | | | T | |
| | | | ONTENTS | |
| | | | IONS | |
| 1. | | | UCTION | |
| 1. | 1.1 | | CAL BACKGROUND | |
| | 1.2 | | G PROFILE | |
| 2. | | | ALE, OBJECTIVES, AND BENEFIT-RISK | ••••• |
| | | | MENT | 10 |
| | 2.1 | | ONALE FOR PERFORMING THE STUDY | |
| | 2.2 | | Y OBJECTIVES | |
| | | | Primary objective | |
| | | 2.2.2 | | |
| | 2.3 | BENE | FIT-RISK ASSESSMENT | |
| 3. | DE | SCRIE | PTION OF DESIGN AND STUDY POPULATION | 11 |
| | 3.1 | | RALL DESIGN AND PLAN | |
| | | 3.1.1 | | |
| | 3.2 | DISCU | USSION OF STUDY DESIGN | |
| | 3.3 | SELE | CTION OF POPULATION | |
| | | 3.3.1 | Main diagnosis for study entry | |
| | | 3.3.2 | Inclusion criteria | |
| | | 3.3.3 | Exclusion criteria | |
| | | 3.3.4 | Removal of patients from therapy or assessments | |
| | | | 3.3.4.1 Removal of individual patients (therapy or assessments) | |
| | | | 3.3.4.2 Discontinuation of the study by the sponsor | |
| 4. | | | <u>IENTS</u> | |
| | 4.1 | | CRIBED TREATMENTS TO BE OBSERVED | |
| | | | Identity of test product(s) and comparator product(s) | |
| | | 4.1.2 | Method of assigning patients to treatment groups | |
| | | | Selection of doses in the study Drug assignment and administration of doses for each patient | |
| | 4.2 | | COMITANT THERAPY, RESTRICTIONS, AND RESCUE | 13 |
| | 4.2 | | TMENT | 13 |
| | | 4.2.1 | Rescue medication, emergency procedures, and additional | 15 |
| | | | treatment(s) | 13 |
| | | 4.2.2 | Restrictions | |
| | | | 4.2.2.1 Restrictions regarding concomitant treatment | |
| | | | 4.2.2.2 Restrictions on diet and life style | |
| 5. | VA | RIABI | LES AND THEIR ASSESSMENT | |
| | | | TY | |

Non-interventional study protocol

BI Trial No.: 1218.104 Doc. No.: UXX-XXX

**** 

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| | | 5.1.1 Endpo | oint(s) of safety | 14 |
|---|---|---|---|---|
| | | 5.1.2 Assess | sment of adverse events | 14 |
| | | 5.1.2.1 | Definitions of adverse events | 14 |
| | | 5.1.2.2 | 2 Adverse event and serious adverse event reporting | 16 |
| | | <b>5.1.3</b> Assess | sment of safety laboratory parameters | 17 |
| | | <b>5.1.4</b> Electr | ocardiogram | 17 |
| | | <b>5.1.5</b> Assess | sment of other safety parameters | 17 |
| | 5.2 | <b>EFFECTIVE</b> | ENESS | 17 |
| | | 5.2.1 Endpo | oint(s) of effectiveness | 17 |
| | | | sment of effectiveness | |
| | 5.3 | | | |
| | 5.4 | <b>APPROPRIA</b> | ATENESS OF MEASUREMENTS | 18 |
| 6. | SU | RVEILLAN | CE PLAN | 19 |
| | 6.1 | VISIT SCHE | EDULE | 19 |
| | 6.2 | | F STUDY PROCEDURES AT SELECTED VISITS | |
| | | | ning and run-in period(s) | |
| | | | ment period(s) | |
| | | | f trial and follow-up period | |
| 7. | ST | | METHODS AND DETERMINATION OF | |
| | | | •••••• | 21 |
| | 7.1 | | AL DESIGN - MODEL | |
| | 7.1 | | ALTERNATIVE HYPOTHESES | |
| | 7.3 | | NALYSES | |
| | 7.5 | | analyses | |
| | | | analyses of effectiveness | |
| | | | analyses of effectiveness | |
| | | | m analyses | |
| | 7.4 | | OF MISSING DATA | |
| | 7.5. | | ATION | |
| | 7.6 | | ATION OF SAMPLE SIZE | |
| 8. | | | CTION, STUDY RECORDS | |
| 0. | | | ROVAL, PATIENT INFORMATION, AND INFORMED | |
| | 0.1 | | | |
| | 8.2 | DATA OHAL | LITY ASSURANCE | 23 |
| | 8.3 | | III ASSURANCE | |
| | 0.5 | | e documents | |
| | | | t access to source data and documents | |
| | | | ge of records | |
| | 8.4 | | LES FOR REPORTING ADVERSE EVENTS | |
| | <b>U.T</b> | | windows | |
| | | | nentation of adverse events and patient narratives | |
| | 8.5 | | T OF CONFIDENTIALITY | |
| | 8.6 | | ON POLICY | |
| 9. | | | | |
| • | | | REFERENCES | |
| | /. | | / INTUITINENDINENDINENDINENDINENDINENDINENDINE | ∠., |

**Boehringer Ingelheim** 

Non-interventional study protocol

BI Trial No.: 1218.104 Doc. No.: UXX-XXX


22 Feb 2017

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| | 9.2 UNPUBLISHED REFERENCES | 26 |
|------------|---------------------------------------|----|
| <b>10.</b> | APPENDICES | 27 |
| | 10.1 ELECTRONIC CASE REPORT FORM | 27 |
| | 10.2 SAE REPORT FORM | 27 |
| | 10.3 PREGNANCY MONITORING FORM | 27 |
| 11. | SUMMARY OF NIS PROTOCOL MODIFICATIONS | 28 |

**Boehringer Ingelheim** 

Non-interventional study protocol 22 Feb 2017

BI Trial No.: 1218.104

Doc. No.: UXX-XXX 

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### **ABBREVIATIONS**

AE Adverse Event

ACR Albumin Creatinine Ratio
ADR Adverse Drug Reaction
CA Competency Authority

CEU Case Entry Unit

CML Clinical Monitor Local CRF Case Report Form

CRO Contract Research Organization

CSO Clinical Safety Officer
DPP-4 Dipeptidyl-peptidase 4

eCRF Electronic Case Report Form

eGFR Estimated Glomerular Filtration Rate

EDC Electronic Data Capture

FU Follow up

FPG Fasting Plasma Glucose

GIP Glucose dependent Insulinotropic Peptide

GLP-1 Glucagon-Like Peptide-1 HbA<sub>1c</sub> Glucosylated Hemoglobin

KFDA Korea Food and Drug Administration KIMS Korea Index of Medical Specialties KPAC Korean Pharmaceutical Affairs Code

KPMA Korea Pharmaceutical Manufacturers Association

KRPIA Korean Research-based Pharmaceutical Industry Association

GCP Good Clinical Practice

ICH International Conference on Harmonisation of Technical

Requirements for Registration of Pharmaceuticals for Human

Use

ID Identification

IEC Independent Ethics Committee IRB Institutional Review Board

MedDRA Medical Dictionary for Drug Regulatory Activities

NCE New Chemical Entity
NIS Non Interventional study
SAE Serious Adverse Event
T2DM Type 2 Diabetes Mellitus
TSAP Trial Statistical Analysis Plan

BI Trial No.: 1218.104 Doc. No.: UXX-XXX 22 Feb 2017

**** 

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 1. INTRODUCTION

#### 1.1 MEDICAL BACKGROUND

Type 2 diabetes mellitus (T2DM) accounts for 90% to 95% of all cases of diabetes and is an increasingly prevalent disease with an estimated 180 million affected people worldwide. Its incidence is expected to double during the next 20 years (R09-4240). In Korea, the prevalence of T2DM patient was 9% in 2010 according to the Diabetes Atlas 4<sup>th</sup> edition from International Diabetes Foundation. Complications induced by hyperglycaemia are currently the most frequent cause of adult-onset loss of vision, renal failure, and non-traumatic lower extremity amputations in the industrialized world. T2DM is also associated with macrovascular complications with a 2- to 4-fold increase in cardiovascular disease risk. The high frequency of complications leads to a significant reduction of life expectancy (R09-4241).

Although several antidiabetic compounds have been developed to improve glucose control and attenuate the metabolic derangements that accompany uncontrolled T2DM, none of these compounds has been able to maintain long-term glycaemic control.

The improved understanding of the incretin effect has contributed to the development of a new class of antidiabetic agents. The incretin effect results from glucagon like peptide-1 (GLP-1) and glucose dependent insulinotropic peptide (GIP), two intestinal peptides that are released in the presence of glucose or nutrients in the gut. GLP-1 stimulates insulin secretion, thereby augmenting glucose-stimulated insulin release. However, there is little risk of hypoglycaemia due to GLP-1 because GLP-1 activity decreases when glucose concentrations fall below 55 milligrams per deciLiter (mg/dL). Normally, GLP-1 is almost instantaneously inactivated by the enzyme DPP-4 that is widely expressed in many tissues including kidney, liver, intestine, lymphocytes and vascular endothelial cells. Therefore, inhibiting DPP-4 would prolong the activity of GLP-1 for stimulating insulin secretion.

Linagliptin is a potent inhibitor of DPP-4 activity and prolongs the half-life of GLP-1. This has been shown in vitro, in various animal models, and in clinical trials. Linagliptin is an orally available compound with a low risk for hypoglycaemic episodes (U04-1767-09).

#### 1.2 DRUG PROFILE

Linagliptin is an orally administered, highly selective DPP-4 inhibitor which is primarily excreted via bile and gut for the treatment of patients with T2DM <sup>2</sup>; its pharmacokinetic and pharmacodynamic profile make it suitable for once-daily dosing (P08-06359, P09-09556).


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 2. RATIONALE, OBJECTIVES, AND BENEFIT-RISK ASSESSMENT

#### 2.1 RATIONALE FOR PERFORMING THE STUDY

According to the local regulations, when a new chemical entity (NCE) is registered, a regulatory non interventional study (rNIS) of an extended period (4 or 6 years) should be conducted. Such rNIS can provide supplementary data to monitor the safety of NCEs in a real-life situation. Data collected in randomised clinical trials with strict inclusion/exclusion criteria and rigorous monitoring schemes have limitations.

This is a prospective, non-interventional, open-label, multi-centre study. It will provide additional safety information of Trajenta in Korean patients with type 2 diabetes mellitus in routine clinical settings.

#### 2.2 STUDY OBJECTIVES

## 2.2.1 Primary objective

The primary objective of this study is to monitor the safety profile of Trajenta in Korean patients with type 2 diabetes mellitus (T2DM) in a routine clinical setting.

## 2.2.2 Secondary objective

The secondary objective of the study is to monitor the effectiveness of Trajenta by evaluating the change from baseline to endpoint in the glycosylated hemoglobin (HbA<sub>1c</sub>), fasting plasma glucose (FPG) of Korean T2DM patients.

#### 2.3 BENEFIT-RISK ASSESSMENT

Patients will be managed according to the local practice guidelines. The choice of treatment will be solely at the discretion of the participating physician. Trajenta will be administered according to the approved label in Korea. Hence there are no additional risks to patients by participating in this rNIS.


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 3. DESCRIPTION OF DESIGN AND STUDY POPULATION

#### 3.1 OVERALL DESIGN AND PLAN

This rNIS is a prospective, non-interventional, open-label, multi-centre study. As per regulation, the re-examination period extends from 14 Sep 2011 until 13 Sep 2017 (6 years). However, active enrollment is to be initiated in 2012 after finalizing the re-imbursement agreement with the authority. Before initiation of the study, any newly reported adverse events collected from other sources such as spontaneous cases, literature cases etc will be closely monitored. The last patient follow up is expected in 2016.

## 3.1.1 Administrative structure of the study

This study will be managed by a project manager of Boehringer Ingelheim Korea. Data management and statistics will be outsourced to a qualified contract research organization (CRO).

#### 3.2 DISCUSSION OF STUDY DESIGN

This is a single arm study with linagliptin.

Loss to follow up

All efforts will be made to minimize loss to follow up, particularly in the tracking of lost patients. To the extent possible, occurrence of adverse event, at minimum, for patients lost to follow up will be obtained. This allows assessing the impact of informative censoring due to treatment discontinuation. Also, patients lost to follow up will be characterized compared to the remaining patients and reason and time point of loss to follow up will be evaluated.

#### Channeling bias

Channeling bias can occur due to preferential prescribing in relation to different risks for the events of interest: e.g., if linagliptin would be more often prescribed to higher risk patients compared to other treatments, higher incidences of outcome events were then expected in the linagliptin group.

## Confounding

As in any observational study, confounding may affect the estimation of associated between drug exposure and outcome of interest and statistical techniques. However, as only major confounders for selected research questions can be captured, residual (unmeasured) confounding may remain.


Doc. No.: UXX-XXX

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 3.3 SELECTION OF POPULATION

A total of 3,000 patients will be enrolled at approximately 80 sites by as many as 100 or more NIS physicians. To minimize the selection bias at the site level, the goal is to have participating centers reflect a balance between general hospitals and clinics for surveillance. The treating physicians will mainly be internists. To minimize the selection bias, consecutive patients from each site who meet inclusion criteria will be enrolled in this study.

## 3.3.1 Main diagnosis for study entry

Patients diagnosed with T2DM will be included.

#### 3.3.2 Inclusion criteria

- Patients who have been started on Trajenta in accordance with the approved label in Korea
- Patients who have signed on the data release consent form

#### 3.3.3 Exclusion criteria

- Patients with previous exposure to Trajenta
- Current participation in clinical trials

#### 3.3.4 Removal of patients from therapy or assessments

#### 3.3.4.1 Removal of individual patients (therapy or assessments)

This section is not applicable.

## 3.3.4.2 Discontinuation of the study by the sponsor

Boehringer Ingelheim Korea reserves the right to discontinue the study overall or at a particular study site at any time for the following reasons:

- 1. Emergence of any effectiveness/safety information that could significantly affect continuation of the study
- 2. Violation of applicable local regulations, the NIS protocol, or the contract by a study site or participating physician, disturbing the appropriate conduct of the study.


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 4. TREATMENTS

#### 4.1 PRESCRIBED TREATMENTS TO BE OBSERVED

## 4.1.1 Identity of test product(s) and comparator product(s)

Trajenta will be prescribed according to the local label and at the discretion of the treating physician. Since this is a non-interventional study, the drug will not be supplied by the sponsor. Furthermore, the sponsor will not cover the expenses related to other medications taken by the patient, interventions, procedures, or diagnostic tests.

## 4.1.2 Method of assigning patients to treatment groups

The choice of treatment is fully at the discretion of the physician and the patient. There is no treatment assignment by a third party.

## 4.1.3 Selection of doses in the study

Linagliptin will be administered 5 mg once a day which is within the authorized label in Korea.

## 4.1.4 Drug assignment and administration of doses for each patient

The physicians indicate doses and timing.

# 4.2 CONCOMITANT THERAPY, RESTRICTIONS, AND RESCUE TREATMENT

The protocol will allow additional drugs considered necessary for the patient's welfare to be prescribed at the discretion of the treating physician. It is required, however, to record the details of all concomitant medication administered to the patient during the course of treatment in eCRF. This includes concomitant therapies started one month prior to Trajenta initiation until the patient completes the final follow-up visit.

## 4.2.1 Rescue medication, emergency procedures, and additional treatment(s)

Please refer to the current local label.

#### 4.2.2 Restrictions

## 4.2.2.1 Restrictions regarding concomitant treatment

Please refer to the current local label.

#### 4.2.2.2 Restrictions on diet and life style

Please refer to the current local label.

BI Trial No.: 1218.104 Doc. No.: UXX-XXX 22 Feb 2017


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 5. VARIABLES AND THEIR ASSESSMENT

#### 5.1 SAFETY

#### 5.1.1 Endpoint(s) of safety

All reported adverse events including hypoglycemic events in patients who take at least one dose of Trajenta will be noted.

Hypoglycemic events include the overall hypoglycemic events, symptomatic hypoglycemia, confirmed hypoglycemia, nocturnal hypoglycemia, and severe hypoglycemia.

Endpoints pertaining to safety will be presented as incidence rates of adverse events and will include:

- adverse events
- unexpected adverse events
- serious adverse events
- drug-related adverse events
- adverse events leading to discontinuation
- adverse events by intensity, outcome of the event, causality

#### 5.1.2 Assessment of adverse events

#### 5.1.2.1 Definitions of adverse events

#### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product. The event does not necessarily have to have a causal relationship with this treatment.

## Serious adverse event

A serious adverse event (SAE) is defined as any AE which results in death, is immediately life-threatening, results in persistent or significant disability / incapacity, requires or prolongs patient hospitalisation, is a congenital anomaly / birth defect, or is to be deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgement which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

Doc. No.: UXX-XXX 

 $Proprietary\ confidential\ information. @\ 2017\ Boehringer\ Ingelheim\ International\ GmbH\ or\ one\ or\ more\ of\ its\ affiliated\ companies.$ 

## Adverse drug reaction

Adverse drug reaction (ADR) refers to any harmful, unintended reaction to the pharmaceutical product of any dose at which a causal relationship with the pharmaceutical product cannot be ruled out.

### Non serious adverse drug reaction

Non serious adverse drug reaction is defined as any ADR which does not meet the SAE criteria.

## Intensity of adverse event

The intensity of the AE should be defined based on the following three categories and according to medical and scientific judgment:

Mild: Transient symptoms which are subjective or objective but no interference with

the patient's daily activities. No change in dosage is needed to continue the

treatment.

Moderate: Marked symptoms with moderate interference with the patient's daily

activities. Reduced dosage or unplanned treatment is necessary for the relief of

adverse events.

Severe: Considerable and unacceptable interference with the patient's daily activities.

Discontinuation of the study drug is required because of significant adverse

events

To ensure that no confusion or misunderstanding of the difference between the terms 'serious' and 'severe' which are not synonymous, it should be noted that SAE does not necessarily correspond to serious or not serious AE to severe ones. All SAEs will be reported regardless of the intensity as mentioned above.

#### Causal relationship of adverse event

Medical judgment will be used to determine the causal relationship, after considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or rechallenge, confounding factors such as concomitant medication, concomitant diseases and relevant history. Assessment of causal relationship will be recorded in the eCRF.

#### Related

- a. Certain: An event occurring in a plausible time relationship to drug administration and that cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug (dechallenge) should be clinically plausible. The event must be definitive pharmacologically or phenomenologically, using a satisfactory rechallenge procedure if necessary.
- b. Probable/Likely: An event with a reasonable time sequence to administration of the drug, unlikely to be attributed to concurrent disease or other drugs or chemicals, and which follows

BI Trial No.: 1218.104 Doc. No.: UXX-XXX

c. No.: UXX-XXX


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

a clinically reasonable response on withdrawal (dechallenge). Rechallenge information is not required to fulfill this definition.

- c. Possible: An event with a reasonable time sequence to administration of the drug, but which could also be explained by concurrent disease or other drugs or chemicals. Information on drug withdrawal may be lacking or unclear.
- d. Conditional/Unclassified: Case of requiring more data or reviewing the additional data for the appropriate assessment
- e. Unassessable/Unclassifiable: Case that it cannot be judged and complemented or confirmed due to the insufficient or contradictory information

#### Unrelated

d. Unlikely: An event with a temporal relationship to drug administration which makes a causal relationship improbable, and in which other drugs, chemicals or underlying disease provide plausible explanations.

Worsening of the underlying disease or other pre-existing conditions

Worsening of the underlying disease or of other pre-existing conditions will be recorded as an (S)AE in the (e)CRF.

Changes in vital signs, ECG, physical examination, and laboratory test results

Changes in vital signs, ECG, physical examination and laboratory test results will be recorded as an (S)AE in the (e)CRF, if they are judged clinically relevant by the NIS physician.

#### 5.1.2.2 Adverse event and serious adverse event reporting

All adverse events occurring from the start of Trajenta treatment up to 7 days after last follow-up visit need to be collected, documented and reported to the sponsor using the AE reporting form of eCRF (Attachment 1). All SAEs must be reported with details of non-serious AEs occurring at the same time, within 24 hours of occurrence via telephone/fax to the Clinical Safety Officer (CSO) of BI Korea using the SAE report form (Attachment2). If any new or further information to these events is available, a follow-up SAE report has to be sent to BI. All SAEs and non-serious AEs must include a causal relationship assessment from the physician.

All other Adverse Events must be reported using eCRFs within 2 weeks to the Sponsor.

## Contact details:

Clinical Safety Officer

Tel: Fax:

Boehringer Ingelheim Non-interventional study protocol BI Trial No.: 1218.104

Doc. No.: UXX-XXX

22 Feb 2017


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Address:

#### Pregnancy

Rarely, patients taking part in regulatory non interventional studies can get pregnant. Once a patient enrolled into the study and exposed to Trajenta becomes pregnant, the NIS physician will stop the drug and report immediately to the sponsor. Drug exposure during pregnancy has to be reported immediately (within 24 hours or next business day, whichever is shorter) to CSO. Furthermore, the details of all the drugs to which the patient exposed at the time of pregnancy will be recorded. The outcome of the pregnancy associated with the drug exposure will be assessed. In the absence of an (S)AE, only the Pregnancy Monitoring Form (Attachment 3) for NIS, not the SAE form is to be completed.

## 5.1.3 Assessment of safety laboratory parameters

This section is not applicable.

### 5.1.4 Electrocardiogram

This section is not applicable.

#### **5.1.5** Assessment of other safety parameters

This section is not applicable.

#### 5.2 EFFECTIVENESS

### **5.2.1** Endpoint(s) of effectiveness

The main effectiveness endpoint in this study is the change from baseline in HbA<sub>1c</sub> after 24 weeks of treatment.

The other effectiveness endpoints are the following:

- Occurrence of treat to target effectiveness response, that is an HbA<sub>1c</sub> under treatment of < 6.5% after 24 weeks of treatment.
- Occurrence of relative effectiveness response (HbA<sub>1c</sub> lowering by at least 0.5% after 24 weeks)
- Change from baseline in fasting plasma glucose (FPG) after 24 weeks of treatment

22 Feb 2017


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### **5.2.2** Assessment of effectiveness

## HbA<sub>1c</sub>:

HbA<sub>1c</sub> should be collected within 1 month prior to baseline and after 12weeks and 24 weeks of treatment.

## Fasting plasma glucose (FPG):

FPG should be collected within 1 month prior to baseline and after 12weeks and 24 weeks of treatment.

## 5.3 OTHER

This section is not applicable.

## 5.4 APPROPRIATENESS OF MEASUREMENTS

This section is not applicable.


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 6. SURVEILLANCE PLAN

#### 6.1 VISIT SCHEDULE

The flow chart at the front of the protocol summarizes the data to be collected at each visit(recommended visit schedule - Visit 2 :  $12\pm2$ weeks/ Visit 3 :  $24\pm2$ weeks). The procedures are further described below.

#### 6.2 DETAILS OF STUDY PROCEDURES AT SELECTED VISITS

#### 6.2.1 Screening and run-in period(s)

This section is not applicable as this is a non-interventional study.

### 6.2.2 Treatment period(s)

As per regulations, enrolled patients will be followed up for 24 week treatment period. There will be a visit window of  $\pm 2$  weeks. To minimize the selection bias at the site level, the goal is to have participating centers reflect a balance between general hospitals and clinics for surveillances.

#### 6.2.2.1 Visit 1 – Baseline Visit

Upon patient enrollment, the following will be recorded on the patient's eCRF.

- Visit date
- Diagnosis: date of the diagnosis of T2DM, family history
- Inclusion / exclusion criteria
- Demographic data: year of birth(age), gender, pregnancy, previous allergy, height, weight, waist circumference, smoking status
- Diabetes mellitus related complication
- Other medical history: history of concomitant disease within 6 months
- Renal Function: record Serum creatinine, eGFR, urin ACR if blood test result is available (collected within the latest 6-month period)
- Effectiveness endpoints : HbA<sub>1c</sub>, FPG (Lab data should be collected within 1month prior to baseline)
- Concomitant anti-hyperglycemic agent: record any anti-hyperglycemic agents have been taken prior to the baseline visit
- Concomitant medications: record all medications have been taken at least once since one month prior to the baseline visit
- Dose of Trajenta given

At Visit 1, the patient will be requested to contact the treating physician in the event of any adverse events noted after initiating Trajenta treatment.

#### 6.2.2.2 Visit 2 (12±2 weeks from Visit 1)

After 12±2 weeks from Visit 1, the patients will return for follow-up. The followings will be noted and recorded in the eCRF:


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Visit date

Doc. No.: UXX-XXX

- Any change of Trajenta given
- Any changes in laboratory tests if there is any lab result which was clinically significant compared to data before Trajenta therapy (This data is collected on the basis of medical need, i.e. independent of the NIS)
- Effectiveness endpoints : HbA<sub>1c</sub>, FPG
- Concomitant anti-hyperglycemic agent including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)
- Concomitant medications including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)
- Any adverse events noted
- Study completion status

#### 6.2.2.3 Visit 3 (24±2 weeks from Visit 1)

After 24±2 weeks from Visit 1, the patients will return for follow-up. The followings will be noted and recorded in the eCRF:

- Visit date
- Any change of Trajenta given
- Any changes in laboratory tests if there is any lab result which was clinically significant compared to data before Trajenta therapy (This data is collected on the basis of medical need, i.e. independent of the NIS)
- Effectiveness endpoints : HbA<sub>1c</sub>, FPG
- Concomitant anti-hyperglycemic agent including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)
- Concomitant medications including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)
- Any adverse events noted
- Study completion status
- NIS physician's electronic signature for data integrity

## 6.2.3 End of trial and follow-up period

Patients with adverse events noted at the final follow-up visit or upon premature discontinuation of Trajenta will be monitored further until the resolution of those adverse events. Alternatively, those patients will be followed up until the NIS physician and sponsor agree that no further follow-up is necessary.


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

Details are provided in the statistical Trial Statistical Analysis Plan (TSAP).

#### 7.1 STATISTICAL DESIGN - MODEL

In this non-interventional study, all statistical analyses will be descriptive. The degree of statistical significance (p-values) and precision (confidence intervals) for the statistical methods used for explorative purposes will be shown. No confirmatory hypotheses are prespecified.

#### 7.2 NULL AND ALTERNATIVE HYPOTHESES

No hypotheses are tested. (See Section 7.1)

#### 7.3 PLANNED ANALYSES

## 7.3.1 Safety analyses

Demographic and baseline characteristics will be summarized descriptively for the entire cohort of eligible patients.

Adverse events (AEs) will be coded according to the latest version of Medical Dictionary for Drug Regulatory Affairs (MedDRA) coding system. Concomitant therapies will be coded according to the latest version of KIMS (Korea Index of Medical Specialties) coding system. The trial database will not be locked until coding is complete.

Safety analyses will be based on all patients treated, i.e. all patients who received at least one dose of Trajenta. However, if data for patients who have been treated with Trajenta beyond the scope of approved label are collected, separate safety analyses will be performed. Safety analyses will be performed based on demographics and baseline characteristics.

Patients lost to follow up will be characterized compared to the remaining patients and reason and time point of loss to follow up will be evaluated.

## 7.3.2 Main analyses of effectiveness

A descriptive analysis of endpoints is planned. For patients treated with Trajenta, the change of HbA<sub>1c</sub> from baseline and last follow-up visit will be calculated. Effectiveness analyses will be performed based on demographics and baseline characteristics.

#### 7.3.3 Other analyses of effectiveness

A descriptive analysis of effectiveness endpoints is planned. For patients treated with Trajenta, the occurrence of treat to target effectiveness response, that is an HbA<sub>1c</sub> under treatment of < 6.5% and relative effectiveness response (HbA<sub>1c</sub> lowering by at least 0.5%)


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

after 24 weeks will be calculated. In addition, the change of FPG from baseline and last follow-up visit will be calculated. Effectiveness analyses will be performed based on demographics and baseline characteristics.

## 7.3.4 Interim analyses

In accordance with local regulation for rNIS, interim analyses are planned biannually for the initial two years and annually thereafter.

#### 7.4 HANDLING OF MISSING DATA

As this is non-interventional study, there are no required investigations and diagnostic procedures (e.g. lab, ultrasound).

Maximum attempt will be made to ensure the completeness of data collection. All available data will be used in the data analysis. There will be no imputation of data to fill the missing values.

#### 7.5. RANDOMISATION

This section is not applicable as this is a non-interventional study.

#### 7.6 DETERMINATION OF SAMPLE SIZE

Sample size of 3,000 patients is based on the requirement of the local regulatory authority (Korean FDA). As per regulation, long-term surveillance is necessary for the indication. Since T2DM is chronic disease, it might be restrictive to collect safety and effectiveness data in short-term (12±2weeks) period, all patients will be enrolled for longer-term (24±2weeks) surveillance.


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 8. DATA PROTECTION, STUDY RECORDS

The International Conference on Harmonization/Harmonized Tripartite Guideline for Good Clinical Practice (ICH/GCP) does not often apply to NIS as most elements are relevant for controlled clinical trials. However, in this NIS, all attempts will be made to adhere, as close as possible, to the standards of ICH/GCP.

The protocol of this regulatory requisite NIS will be submitted to the Korea Food and Drug Administration (KFDA) for notification. It is not a local requirement in Korea to obtain Institutional Review Board (IRB) approval for the conduct of regulatory requisite NIS. However, the protocol of this NIS will be submitted to IRBs whenever required or requested by these institutions. This study will be conducted in accordance with the Standards for Reexamination of New Medicines notified by KFDA, Korean Pharmaceutical Affairs Code (KPAC), Enforcement Regulation of KPAC and other applicable local laws and industry code (including but not limited to the Regulations on Fair Competition in the Trade of Medicines of KPMA and KRPIA).

Boehringer Ingelheim Korea will submit periodic reports during re-examination period, and the final report to KFDA upon study completion. The periodic report for the final year will be substituted with the final report. When required, the interim reports and the final report will be submitted to the IRBs as well.

# 8.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This study will be initiated only after all required legal documentation has been reviewed and approved by the respective IRB/IEC and the competent authority (CA) according to the local regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the study, written data release consent form shall be obtained from each patient (or the patient's legally accepted representative). Each signature must be personally dated by each signatory and the data release consent and any additional patient-information form retained by the NIS physician as part of the trial records. A signed copy of the data release consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

The patient must be informed that his/her personal study-related data will be used by Boehringer Ingelheim Korea in accordance with the local data protection law. The level of disclosure shall also be explained to the patient.

The patient shall be informed that his/her medical records may be examined by authorised monitors (MPMs) or Clinical Quality Assurance auditors appointed by sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 8.2 DATA QUALITY ASSURANCE

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by IRBs/IECs or by regulatory authorities. The quality assurance auditor will have access to all medical records, the participating physician's study-related files and correspondence, and the data release agreement documentation of this study.

#### 8.3 RECORDS

Doc. No.: UXX-XXX

All of the clinical data will be captured via a web-based EDC (Electronic Data Capture) System. The site staff will enter and edit the data via a secure network, with secure access features (username, password and secure identification – an electronic password system). A complete electronic audit trail will be maintained. The treating physician will approve the data using an electronic signature.

Patients will not be identified on the eCRF by name. Appropriate coded identification (i.e., patient number) will be used. The treating physician will make a separate confidential record of these details (patient identification code list) to permit identification of all patients enrolled in this study in case follow-up is required. Likewise, any supporting documentation will be redacted of any patient identifying information, and the patient ID number clearly written on the documents.

#### **8.3.1** Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents will be filed at the treating physician's site.

It is necessary that the data entered in the eCRFs that are transcribed from the source documents are consistent with the source documents or the discrepancies need to be explained. The treating physician may need to request previous medical records, transfer records, and current medical records.

#### 8.3.2 Direct access to source data and documents

The NIS physician / site will permit study-related monitoring, audits and regulatory inspection, providing direct access to all related source data/documents. All source documents including eCRFs will be made available for review by sponsor's Medical Project Manager (MPM) or designees and inspection by health authorities (e.g., KFDA). The MPM and auditor may review all eCRFs, and written data release agreements. The accuracy of the data will be verified by reviewing the documents described in Section 8.3.1.

## 8.3.3 Storage of records

The NIS physician and the site are jointly responsible for maintaining essential study documents for 3 years after completion of the study (defined as termination date of reexamination period) by the Pharmaceutical Affairs Law and shall take measures to prevent accidental or premature destruction of these documents.


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 8.4 PROCEDURES FOR REPORTING ADVERSE EVENTS

#### **8.4.1** Time windows

Doc. No.: UXX-XXX

All AEs, serious and non-serious, occurring during the course of the rNIS will be collected, documented and reported to the sponsor by the investigator on the appropriate eCRF. Reporting will be done according to the specific definitions and instructions detailed in the 'Adverse Event Reporting' section of the site materials (that include all necessary documents, the protocol, instructions for conducting rNIS, the package insert etc.).

The investigator has the responsibility to report AEs during the specified observational phase.

Any SAE, whether or not considered related to Trajenta tablets, or whether or not Trajenta tablets has been administered, must be reported immediately via eCRF.

## 8.4.2 Documentation of adverse events and patient narratives

Expedited reporting of serious adverse events, e.g. suspected unexpected serious adverse reactions (SUSARs) to health authorities and IECs/IRBs, will be done according to the local regulatory requirements.

For each AE, the investigator will provide the onset, end, intensity, outcome, seriousness and action taken with Trajenta tablets. The investigator will determine the relationship of Trajenta tablets to all AEs as defined in the 'Adverse Event Reporting' section of the physician binder.

#### 8.5 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this study will be considered confidential and disclosure to third parties will be prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Treatment data will be made available to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated from the study will be made available for inspection on request by the participating physicians, the sponsor and/or its representatives and/or designees, by the IRBs/IECs and the regulatory authorities.

#### **8.6 PUBLICATION POLICY**

Boehringer Ingelheim, to the best of their ability will support the process of free exchange of relevant scientific information. Any publication of the result of this NIS study must be consistent with the Boehringer Ingelheim publication policy.


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 9. REFERENCES

Doc. No.: UXX-XXX

#### 9.1 PUBLISHED REFERENCES

- R09-4240 World Health Organization. Diabetes. http://www.who.int/mediacentre/factsheets/fs312/en/; (WHO Fact sheet; no 312) 2008.
- R09-4241 Haffner SM, Letho S, Rönnemaa T, Pyörälä K, Laakso M. Mortality from coronary heart disease in subjects with type 2 diabetes and in non-diabetic subjects with and without prior myocardial infarction. N. Engl. J. Med. 1998; 339 (4): 229-234.
- P08-06359 Thomas L et al., (R)-8-(3-amino-piperidin-1-yl)-7-but-2-ynyl-3-methyl-1-(4-methyl-quinazolin-2-ylmethyl)-3,7-dihydro-purine-2,6-dione (BI 1356), a novel xanthine-based dipeptidyl peptidase 4 inhibitor, has a superior potency and longer duration of action compared with other dipeptidyl peptidase-4 inhibitors. J Pharmacol Exp Ther. 2008; 325: 175–82
- P09-09556 Graefe-Mody EU et al., Evaluation of the potential for steady-state pharmacokinetic and pharmacodynamic interactions between the DPP-4 inhibitor linagliptin and metformin in healthy subjects. Curr Med Res Opin. 2009; 25: 1963–72

#### 9.2 UNPUBLISHED REFERENCES

U04-1767-09 Linagliptin Investigator's Brochure. Version 9. 10 Dec 2010.

- International Diabetes Federation.
  http://www.idf.org/diabetesatlas/
  Prevalence extimates of diabetes mellitus, 2010, The Diabetes Atlas 4th edition
- et al., Safety, tolerability, pharmacokinetics, and pharmacodynamics of single oral doses of BI 1356, an inhibitor of dipeptidyl peptidase 4, in healthy male volunteers. J Clin Pharmacol. 2008; 48: 1171–8
- 3 Treatment Guideline for Diabetes 2011, Korean Diabetes Association

BI Trial No.: 1218.104 Doc. No.: UXX-XXX


22 Feb 2017

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 10. APPENDICES

## 10.1 ELECTRONIC CASE REPORT FORM

See the Attachment 1.

## 10.2 SAE REPORT FORM

See the Attachment 2.

## 10.3 PREGNANCY MONITORING FORM

See the Attachment 3.

22 Feb 2017

Doc. No.: UXX-XXX 

Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 11. SUMMARY OF NIS PROTOCOL MODIFICATIONS

**Summary of Modifications Sheet (SOMS)** 

| Number of Protocol modification | 1 |
|---|---|
| D ( CD ( ) 1°C ( | |
| Date of Protocol modification | 13 Sep 2012 |
| BI Trial number | |
| | 1218.104 |
| BI Product(s) | |
| | Trajenta |
| Title of protocol | A regulatory requirement non interventional study to monitor the safety and effectiveness of Trajenta (Linagliptin, 5 mg, q.d) in Korean patients with type 2 diabetes mellitus |
| | SELINA study |
| To be implemented only after | |
| approval of the | |
| IRB/IEC/Competent Authorities | |
| To be implemented immediately | <u> </u> |
| in order to eliminate hazard – | |
| IRB / IEC / Competent Authority | |
| to be notified of change with | |
| request for approval | |
| Can be implemented without | |
| IRB/IEC/ Competent Authority | |
| approval as changes involve | |
| logistical or administrative | |
| aspects only | |
| Section to be changed | Refer to amendment table |
| Description of change | |
| Rationale for change | |


Proprietary confidential information. © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| Number of Protocol modification | 2 |
|---|---|
| Date of Protocol modification | 22 Feb 2017 |
| BI Trial number | 1218.104 |
| BI Product(s) | Trajenta |
| Title of protocol | A regulatory requirement non interventional study to monitor the safety and effectiveness of Trajenta (Linagliptin, 5 mg, q.d) in Korean patients with type 2 diabetes mellitus SELINA study |
| To be implemented only after | |
| approval of the | |
| IRB/IEC/Competent Authorities | |
| To be implemented immediately | |
| in order to eliminate hazard – | |
| IRB / IEC / Competent Authority | |
| to be notified of change with | |
| request for approval | |
| Can be implemented without | |
| IRB/IEC/ Competent Authority | |
| approval as changes involve | |
| logistical or administrative | |
| aspects only | |
| uspecto only | 1 |
| Section to be changed | Refer to amendment table |
| Description of change | Telef to afficient table |
| Rationale for change | $\dashv$ |
| Kationale for change | |